

## T.C. GAZI UNIVERSITY RECTORATE Ethics Committee

Number :E-77082166-604.01.02-487579

19.10.2022

Subject : Evaluation and Approval

Dear Assoc. Prof. Dr. Zait Burak AKTUĞ Nigde Ömer Halisdemir University Faculty of Sports Sciences

The research proposal titled "The Effects of Low-Intensity Cycling Exercises Combined with the Blood Flow Restriction Method on MaxVO<sub>2</sub>, Muscle Strength, and Muscle Thickness," submitted by the research group consisting of Zait Burak AKTUĞ, Serkan İBİŞ, Cengiz AKARÇEŞME, Hasan AKA, Bökebatur Ahmet Raşit MENDİ, Necdet Eray PİŞKİN, and Gönül YAVUZ, was reviewed during our Committee's meeting No. 16 held on 04.10.2022.

It was unanimously decided that there is no ethical objection to conducting your study, provided that the necessary permissions are obtained from the institutions where the research is to be conducted. The signature list related to this decision is attached.

Sincerely,

Research Code No: 2022 - 961

Prof. Dr. Fazlı POLAT Vice Rektor

Attachment: 1 List

This document has been signed with a secure electronic signature.

Document Verification Code: BSCEFUUBH2

Adress: https://www.turkiye.gov.tr/gazi-universitesi-ebys

For information: Ayfer Çekmez General Documents Officer Phone Number: 202 38 81



## GAZI UNIVERSITY ETHICS COMMITE PARTICIPANT LIST MEETING DATE: 04.10.2022 MEETING NUMBER: 16 NAME-SURNAME SIGNATURE Prof. Dr. İsmail KARAKAYA MODERATOR